CLINICAL TRIAL: NCT01291732
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses (12.5 mg, 50 mg, 200 mg) of BI 135585 XX (Tablet) in Chinese and Japanese Healthy Male Volunteers (Randomised, Double-blind,Placebo-controlled Within Dose Groups)
Brief Title: Single Rising Dose Study of BI 135585 XX in Health Asian Male Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1283.5
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Healthy

ARMS (2):
- BI 135585 XX (Experimental): single dose of BI 135585
  Interventions: Drug: BI 135585 XX
- matching placebo (Placebo Comparator): single dose of matching placebo
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Matching placebo — single dose of matching placebo
  Arms: matching placebo
Drug: BI 135585 XX — single dose of low, medium or high dose of BI 135585 XX
  Arms: BI 135585 XX

SUMMARY:
The Aim of the study is to evaluate safety, tolerability, pharmacokinetics and pharmacodynamics in Asian healthy males administered a single dose of BI 135585.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male volunteers,
2. Chinese or Japanese ethnicity

Exclusion criteria:

1. Any finding of the medical examination (including blood pressure (BP), pulse rate (PR) and electrocardiogram (ECG)) deviating from normal and of clinical relevance according to the investigators medical judgement
2. Any evidence of a clinically relevant concomitant disease
3. Intake of drugs with long half life (>24 hour) within at least one month or less than 10 half-lives of the respective drug prior to administration

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Changes in Vital signs (blood pressure (BP), pulse rate (PR), respiratory rate(RR)) | up to 21 days
Changes in 12-lead ECG (electrocardiogram) | up to 21 days
Changes in Clinical laboratory tests (haematology, clinical chemistry and urinalysis) | up to 21 days
Occurrence of Adverse events | up to 21 days

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | 10 days
Tmax (maximum measured concentration of the analyte in plasma) | 10 days
AUC0-8 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1283.5.82001 Boehringer Ingelheim Investigational Site, Seoul, South Korea